CLINICAL TRIAL: NCT00040521
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of Orally Administered Recombinant Human Interleukin-11 (rhIL-11) for the Treatment of Patients With Active Crohn's Disease
Brief Title: Study Evaluating rhIL-11 in Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 3067K5-208; B2491021 (Other: Pfizer)
Record Dates: First submitted 2002-06-27; First posted 2002-06-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2005-09

CONDITIONS: Crohn Disease; Inflammatory Bowel Disease
Keywords: Crohn's Disease; Active Crohns Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Interleukin-11; oprelvekin

INTERVENTIONS:
Drug: Recombinant Human Interleukin-11 (rhIL-11)

SUMMARY:
The purpose of this study is to assess the activity of multiple doses of oral rhIL-11 in patients with active Crohn's disease (Crohn's Disease Activity Index [CDAI] score from 220-400).

ELIGIBILITY:
Inclusion Criteria:

* Documented, signed and dated informed consent to participate in this trial prior to any study related procedures being performed.
* Men and women age 16 years and over.
* Diagnosis of Crohn's disease for at least 6 months that has been appropriately documented and confirmed by radiological studies, endoscopy (with histological examination preferred), or surgical pathology (Patients with a diagnosis of Crohn's disease for less than 6 months may be included if the diagnosis is confirmed by a biopsy characteristic of Crohn's disease)

Exclusion Criteria:

Use of the following medications within the specified time period prior to randomization:

* Nonsteroidal anti-inflammatory drugs (NSAIDs; including Cyclooxygenase-2 [COX-2] inhibitors and >500 mg/day acetylsalicylic acid)
* Codeine-containing compounds
* Corticosteroid enemas

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — clinicaltrialinfo@wyeth.com
Locations (2):
- United States (2):
  - Arvada, Colorado
  - Chapel Hill, North Carolina